CLINICAL TRIAL: NCT00488540
Title: Is Paracetamol an Effective Treatment for Chronic Moderate Pain in the Newborn After Operative Vaginal Delivery?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Neonatology and Obstetrics, University Hospital Inselspital Berne (Unknown); University Hospital, Zürich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 291/06
Record Dates: First submitted 2007-06-19; First posted 2007-06-20 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Pain
Keywords: newborn; infant; pain; acetaminophen; paracetamol; mode of delivery; vacuum extraction; forceps extraction; cesarean section; EDIN scale; Bernese Pain Scale for Neonates; pain after different modes of delivery in newborn infants; efficacy of acetaminophen as analgesia for newborn infants
MeSH Terms: conditions — Pain | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paracetamol (Acetaminophen) (Active Comparator): Paracetamol (Acetaminophen) given at 2 and 8 hours post birth, measurement of EDIN-Score on day one of life, measurement of stress response after Guthrie-test on day 4 of life.
  Interventions: Drug: Paracetamol
- Placebo (Placebo Comparator): Placebo given at 2 and 8 hours post birth, measurement of EDIN-Score on day one of life, measurement of stress response after Guthrie-test on day 4 of life.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Paracetamol — Suppository
  Other Names: Acetaminophen
  Arms: Paracetamol (Acetaminophen)
Drug: Placebos — Suppository
  Arms: Placebo

SUMMARY:
There are many reasons for using a vacuum apparatus or forceps to assist in delivering a baby. The traction and pressure on the baby's head due to the vacuum apparatus or forceps may cause pain and discomfort for some time after the delivery. To date, the pain experienced by the newborn and the potential beneficial effects of pain medications after vacuum or forceps deliveries have not been systematically studied. It is possible that administration of paracetamol suppositories to the newborn may be helpful in these situations, since this medication is known to ameliorate pain in older children and adults.

DETAILED DESCRIPTION:
How will this study be conducted?

The study will be conducted in the Women's University Hospital of Basel, the Women's University Hospital of Zurich and the Women's University Hospital of Bern. Newborn infants born with the aid of a vacuum or forceps will be included, with the explicit permission of their parents. The children will receive a rectal suppository, which will be prepared by the pharmacy at the Women's University Hospital of Basel, at two and eight hours of postnatal age. These children will receive either paracetamol or a placebo, which will be randomly assigned. The doctors, the midwives, nurses and other people involved in the care of the child will not know which medication had been given. Only the pharmacy has access to this information, which can be obtained only in emergency situations. The child will be regularly monitored for signs of pain or discomfort.

In Switzerland, all newborn babies are tested at three days of age for thyroid and other rare but treatable diseases by taking a blood sample from the heel. Newborns that participate in this study will be observed after this blood draw to see how long they show signs of pain or discomfort. In addition, sputum tests before and after the blood draw will be taken in order to measure the level of cortisone (a measurement of stress).

What measures will be performed?

* Two suppositories, either with or without paracetamol, will be administered (only to children in the study group, that is, those that were born with the aid of a vacuum or forceps).
* On the first day of life, at 2, 4, 8, 12 and 24 hours after delivery, a midwife or nurse will examine the newborn (EDIN scale) and determine if he or she has pain, and if so, will indicate how strong the pain appears to be.
* On the fourth day of life, at the same time that the standard blood screening tests for metabolic diseases are performed, a saliva test to identify the stress hormone cortisol will be taken before and after the blood tests and the pain reaction will be measured. The length of time that the child cries after the blood test has been performed will be observed and filmed, in order to more accurately determine the duration of the crying. This film will be destroyed after the study has been completed.
* As with all other newborns, we will give the child a small amount of sugar solution before taking the blood sample to reduce the pain. The efficacy of this measure has been well documented.

No child will have additional blood tests outside of the routinely performed screening tests through participation in this study.

In order to determine whether babies born by caesarean section or without any assistance through instruments such as vacuum or forceps experience less pain and have a less dramatic stress reaction, we will enroll also children, who were born without the aid of one of these instruments, for observation in this study. They will not receive any medication.

ELIGIBILITY:
Inclusion Criteria:

* Newborns after vacuum or forceps extraction for paracetamol or placebo
* Newborns after vaginal delivery or cesarean section as observational group
* Gestational age at or above 35 weeks
* Birthweight above 2000g
* Signed informed consent of parents

Exclusion Criteria:

* Multiples
* Fetal malformation
* Systemic opiates within 24 hours before birth
* Ambulatory birth (mother and child leave the hospital a few hours after birth)

Ages: 30 Minutes to 1 Hour | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 280 (Estimated)
Dates: Start 2007-06; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Measurement of pain reaction using the EDIN scale on the first day of life and evaluation of the stress-reaction after the Guthrie test with duration of crying, saliva cortisol and "Bernese Pain Scale for Neonates"

SECONDARY OUTCOMES:
Validation of the Bernese Pain Scale for Neonates and the EDIN scale. Comparison between different types of vacuum extractors in view of neonatal pain. Comparison of different modes of delivery in view of neonatal pain and stress-reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Hösli, Prof. Dr. MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (3):
- Switzerland (3):
  - University Hospital Basel, Basel, Canton of Basel-City
  - Neonatology and Obstetrics, University Hospital Inselspital Berne, Bern
  - Neonatology and Obstetrics, University Hospital Zurich, Zurich

REFERENCES:
- [Background] Debillon T, Zupan V, Ravault N, Magny JF, Dehan M. Development and initial validation of the EDIN scale, a new tool for assessing prolonged pain in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2001 Jul;85(1):F36-41. doi: 10.1136/fn.85.1.f36. PMID 11420320
- [Background] Cignacco E, Mueller R, Hamers JP, Gessler P. Pain assessment in the neonate using the Bernese Pain Scale for Neonates. Early Hum Dev. 2004 Jul;78(2):125-31. doi: 10.1016/j.earlhumdev.2004.04.001. PMID 15223117
- [Result] Schuller C, Kanel N, Muller O, Kind AB, Tinner EM, Hosli I, Zimmermann R, Surbek D. Stress and pain response of neonates after spontaneous birth and vacuum-assisted and cesarean delivery. Am J Obstet Gynecol. 2012 Nov;207(5):416.e1-6. doi: 10.1016/j.ajog.2012.08.024. Epub 2012 Aug 17. PMID 22959831
- [Result] Tinner EM, Hoesli I, Jost K, Schobi N, Ulrich Megged Y, Burkhardt T, Krafft A, Bucher HU, Surbek D, Nelle M, Buhrer C. Rectal paracetamol in newborn infants after assisted vaginal delivery may increase pain response. J Pediatr. 2013 Jan;162(1):62-6. doi: 10.1016/j.jpeds.2012.06.020. Epub 2012 Jul 17. PMID 22809664
- [Result] Huhn EA, Visca E, Vogt DR, von Felten S, Tinner Oehler EM, Buhrer C, Surbek D, Zimmermann R, Hoesli I. Decreased neonatal pain response after vaginal-operative delivery with Kiwi OmniCup versus metal ventouse. BMC Pregnancy Childbirth. 2017 Jan 31;17(1):47. doi: 10.1186/s12884-017-1231-x. PMID 28143599